CLINICAL TRIAL: NCT00139685
Title: Depo-Provera: Evaluation of Bone Mineral Density and Total Body Calcium in Adolescent DP 150 CI Users and Matched Controls
Brief Title: Depo-Provera: Bone Mineral Density and Total Body Calcium in Adolescent DP150CI Users and Non-Hormonal Contraception
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Z54000261; NCT00264836 (obsolete NCT alias)
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Contraception; Bone Density

INTERVENTIONS:
Drug: Depo-Provera Contraceptive Injection - DP150CI

SUMMARY:
To evaluate and compare Bone Mineral Density (BMD) in adolescent Depo-Provera Contraceptive Injection (DP150CI) users during depo medroxyprogesterone acetate (DMPA) therapy and following discontinuation of DMPA. Another group electing non-hormonal contraception or abstinence will be recruited as a reference population, across all study sites. The primary variable is BMD, measured by Dual Energy X-ray Absorptiometry (DXA). Secondary variables are: Total Body Composition& Total Body Calcium (TBC), measured by Dual Energy X-ray Absorptiometry (DXA), and surrogate biologic BMD markers. Safety will be evaluated by adverse event reporting, laboratory evaluations, pregnancies, weight and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent females who have had any menses in the 6 months prior to enrollment
* Must have a negative pregnancy test

Exclusion Criteria:

* Concomitant medication exclusion use of bone modifying agents, glucocorticoids, heparin, and anticonvulsants
* Screening Spinal BMD with z score not greater than -2 of matched young normals

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350
Dates: Start 1998-04; Primary Completion 2006-08 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Changes in Bone Mineral Density in adolescent Depo-Provera Contraceptive
Injection (DP150CI) users will be evaluated and compared during depo
medroxyprogesterone acetate (DMPA) therapy and following discontinuation of
DMPA.Another group electing non-hormonal contraception or abstinence is
recruited as a reference population, across all study sites.

SECONDARY OUTCOMES:
Secondary variables are: Total Body Composition & Total Body Calcium (TBC),
measured by Dual Energy X-ray Absorptiometry (DXA)Surrogate biologic BMD
markers

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Norfolk, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=Z54000261&StudyName=Depo%2DProvera%3A+Evaluation+of+BMDensity+and+Total+Body+Ca+Adolescent+DP150CI+Users+and+Non%2Dhormonal+Contraception